CLINICAL TRIAL: NCT00842088
Title: A Randomized, Blinded, Placebo-controlled, Dose Escalation Study to Evaluate the Safety, Tolerability and Pharmacokinetics of HQK-1001 in Subjects With Sickle Cell Disease
Brief Title: Phase 1/2 Study to Evaluate the Safety, Tolerability and Pharmacokinetics of HQK-1001 Administered Daily in Patients With Sickle Cell Disease
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: HemaQuest Pharmaceuticals Inc. (Industry)
Responsible Party: Susan Perrine, M.D., HemaQuest Pharmaceuticals, Inc.
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HQP 2008-004
Record Dates: First submitted 2009-02-11; First posted 2009-02-12 (Estimated); Last update posted 2011-08-01 (Estimated); Status verified 2011-07

CONDITIONS: Sickle Cell Disease
MeSH Terms: conditions — Anemia, Sickle Cell | interventions — 2,2-dimethylbutyric acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Active (Experimental)
  Interventions: Drug: HQK-1001
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Placebo — Matching placebo capsule. Administered orally once a day on dosing days.
  Arms: Placebo
Drug: HQK-1001 — HQK-1001 capsules. 10 mg/kg, 20 mg/kg or 30 mg/kg administered once a day on dosing days.
  Arms: Active

SUMMARY:
The purpose of this study is to assess the safety and tolerability of HQK-1001 administered for a total of 12 weeks (with one dosing break) in subjects with sickle cell disease.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of SCD or sickle beta thalassemia (excluding Hemoglobin C)
* Between 12 and 60 years of age, inclusive
* At least one episode of a SCD-related crisis or complication (e.g., vaso-occlusive crisis, acute chest syndrome, priapism) per year for an average of 3 years or one episode of acute chest syndrome over the prior 5 years
* Screening (untransfused) HbF level >/= 2% as analyzed by a central laboratory
* If receiving hydroxyurea therapy, must be receiving a stable dose for at least 6 months
* Able and willing to give informed consent
* If female, must have a negative serum pregnancy test within 7 days of dosing
* If female, must not be of childbearing potential defined as post-menopausal by at least 2 years or surgically sterile, or must agree to use a medically accepted form of contraception throughout the study
* If the sexual partner of a male subject is a WCBP, she must agree to use a medically accepted form of birth control for themselves or their partner throughout the study
* In the view of the Investigator, able to comply with necessary study procedures

Exclusion Criteria:

* Red blood cell (RBC) transfusion within 3 months prior to beginning study medication
* Participation in a regular blood transfusion program
* More than 4 hospitalizations for acute sickle cell-related events in the previous 12 months
* An acute vaso-occlusive event within 3 weeks prior to receiving first dose of study medication
* Pulmonary hypertension requiring oxygen
* QTc > 450 msec on screening
* Alanine transaminase (ALT) > 3X upper limit of normal (ULN)
* Creatinine phosphokinase (CPK) > 20% above the ULN
* Serum creatinine >1.2 mg/dL
* An acute illness (e.g., febrile, gastrointestinal [GI], respiratory) within 72 hours prior to receiving first dose of study medication
* History of syncope, clinically significant dysrhythmias or resuscitation from sudden death
* Chronic opiate use which, in the view of the Investigator, could confound evaluation of an investigational drug
* Current abuse of alcohol or drugs
* Received another investigational agent within 4 weeks, or 5 half-lives, whichever is longer, prior to administration of study medication
* Currently pregnant or breast feeding a child
* Known infection with HIV-1
* Infection with hepatitis B or hepatitis C such that patients are currently on therapy or will be placed on therapy during the trial

Ages: 12 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 24 (Actual)
Dates: Start 2009-03; Primary Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Safety as assessed by (1) adverse events (2) laboratory values (3) vital signs, and (4) physical exam. | 126 days

SECONDARY OUTCOMES:
Pharmacokinetics assessed by plasma drug concentration levels. | Days 0, 6, 69 and 97 post first dose
Pharmacodynamics assessed by red blood cell production and induction of fetal hemoglobin. | Every 2 weeks through Day 126 post first dose

CONTACTS AND LOCATIONS:
Overall Officials: Susan Perrine, M.D., Study Director — HemaQuest Pharmaceuticals
Locations (9):
- United States (8):
  - Trialogic Research, Madison, Alabama
  - Children's Hospital and Research Center at Oakland, Oakland, California
  - Century Clinical Research, Inc., Daytona Beach, Florida
  - Medical College of Georgia, Augusta, Georgia
  - University of Illinois at Chicago, Chicago, Illinois
  - Johns Hopkins School of Medicine, Baltimore, Maryland
  - UNC Comprehensive Sickle Cell Program, Chapel Hill, North Carolina
  - Texas Children's Cancer Center and Hematology Service, Houston, Texas
- University of the West Indies, Mona, Kingston, Mona, Jamaica

REFERENCES:
- [Derived] Kutlar A, Ataga K, Reid M, Vichinsky EP, Neumayr L, Blair-Britt L, Labotka R, Glass J, Keefer JR, Wargin WA, Berenson R, Perrine SP. A phase 1/2 trial of HQK-1001, an oral fetal globin inducer, in sickle cell disease. Am J Hematol. 2012 Nov;87(11):1017-21. doi: 10.1002/ajh.23306. Epub 2012 Aug 7. PMID 22887019